CLINICAL TRIAL: NCT05500625
Title: Endoscopic Ultrasound-guided Coil With Cyanoacrylate Injection Versus Balloon-Occluded Retrograde Transvenous Obliteration in Managing Patients With Gastric Varices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Mohammed Mahrous Sayed, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUSCCIBRTOMPGV
Record Dates: First submitted 2022-07-29; First posted 2022-08-15 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Gastric Varix
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-guided coil embolization combined with endoscopic cyanoacrylate injection (Experimental)
  Interventions: Procedure: Endoscopic ultrasound-guided coil embolization combined with endoscopic cyanoacrylate injection
- Ballon-occluded retrograde transvenous obliteration (Experimental)
  Interventions: Procedure: Ballon-occluded retrograde transvenous obliteration

INTERVENTIONS:
Procedure: Endoscopic ultrasound-guided coil embolization combined with endoscopic cyanoacrylate injection — Standard diagnostic endoscopy will be done and Fundal varices will be assessed. EUS procedures will be performed using linear endoscope under general anesthesia. Use EUS to assess the anatomy of gastric varices, observe the blood flow, scan the portal venous system, left renal vein, confirm the location of the shunt, and measure the diameter of the shunt. Puncture the gastric fundal variceal vein at the lower esophagus near the cardia and place the coil into the shunt and immediately inject with sclerosant and cyanoacrylate under the guidance of EUS using a sandwich method (cyanoacrylate, sclerosant and cyanoacrylate) via endoscope. Use color Doppler ultrasound to observe the blood flow in the variceal veins to evaluate the embolization effect.
  Other Names: EUS-guided coil embolization combined with endoscopic cyanoacrylate injection
  Arms: EUS-guided coil embolization combined with endoscopic cyanoacrylate injection
Procedure: Ballon-occluded retrograde transvenous obliteration — A balloon occlusion catheter will be inserted into the venous end of the gastro-renal or gastro-caval shunt via the right femoral vein or internal jugular vein. Balloon-occluded retrograde venogram will be done to evaluate degree of retrograde filling of the gastric varices and presence of collateral veins. Any significant large collateral veins seen will be occluded with coils using microcatheter to prevent leakage of the sclerosant into the systemic circulation. Then, sclerosant agent (ethanol-amine oleate, Sodium tetradecyl sulphate, or polidocanol) will be injected into the portosystemic shunt till complete filling of the gastric varices and part of the feeding veins. Finally, the balloon left in place for 2-12 hours then gradually will be deflated when complete occlusion of blood flow of the target shunt is achieved.
  Other Names: BRTO
  Arms: Ballon-occluded retrograde transvenous obliteration

SUMMARY:
Gastrointestinal bleeding is a common complication of liver cirrhosis which caused by esophageal and gastric varices. The risk of bleeding from gastric varices is relatively low. However, the bleeding is usually significant and severe.

Current guidelines recommend endoscopic glue injection as the first line of treatment for gastric variceal bleeding.

Although this technique has been shown to be effective, it is associated with many severe adverse events including systemic embolization, fever, chest pain, and even death. The rate of hemostasis has been reported to be as high as 91-100% but the rebleeding rate from gastric varices still present.

Endoscopic ultrasound (EUS) guided therapy has recently been introduced as a more effective and safer option than endoscopic therapy for gastric varices. EUS-guided therapy includes EUS guided Cyanoacrylate injection alone or in combination with EUS-guided coiling. It offers the advantage of directly visualizing the varices and delivering targeted therapy.

A standard endoscopic examination only allows the evaluation of superficial varices. The use of Endoscopic ultrasound facilitates evaluation of peri-gastric and perforating vessels, which are directly involved in variceal development. EUS also facilitates accurate placement of the coil and preserves the naturally formed splenorenal shunt.

Balloon-occluded retrograde transvenous obliteration(BRTO) has been reported to achieve satisfactory bleeding control rates for isolated gastric varices with High hemostasis rates and low rebleeding rate.

Despite all these promising results, there are scarce studies describing and comparing the efficacy of EUS-guided therapy and BRTO in patients with gastric varices. Further prospective comparative studies are needed.

ELIGIBILITY:
Inclusion Criteria:

• Presence of fundal gastric varices either: High risk for rupture; diagnosed by upper endoscopy i.e. large size or presence of red color spot.

Bleeding varices; diagnosed by upper endoscopy with good hemostasis achieved with endoscopic treatment.

Bleeding varices; diagnosed by upper endoscopy but hemostasis could not be achieved with endoscopic treatment.

* Fundal gastric varices with Presence of contraindication for TIPS such as repeated attacks of hepatic encephalopathy due to Portosystemic shunt, Model of End Stage Liver disease score (MELD) >18.
* Fundal varices with catheterizable portosystemic shunt such as gastrorenal shunt or gastrocaval shunt.

Exclusion Criteria:

* Complete portal vein thrombosis
* Splenic vein thrombosis
* Intractable ascites (TIPS is better)
* Uncontrolled esophageal varices (high risk for bleeding) and TIPS is better

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-08-30 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Gastric varices bleeding control | 7 days
  Teatment using EUS- guided coil with cyanoacrylate injection in group of patients and other group treatment using Balloon-Occluded Retrograde Transvenous Obliteration Gastric varices bleeding control within 1 week The parameter will be assesed is incidence of bleeding after the procedure number of attacks of haematemsis and melena)
Time of procedure | 1 day
  Time of the whole procedure of EUS and BRTO

REFERENCES:
- [Background] Boregowda U, Umapathy C, Halim N, Desai M, Nanjappa A, Arekapudi S, Theethira T, Wong H, Roytman M, Saligram S. Update on the management of gastrointestinal varices. World J Gastrointest Pharmacol Ther. 2019 Jan 21;10(1):1-21. doi: 10.4292/wjgpt.v10.i1.1. PMID 30697445
- [Background] Baig M, Ramchandani M, Puli SR. Safety and efficacy of endoscopic ultrasound-guided combination therapy for treatment of gastric varices: a systematic review and meta-analysis. Clin J Gastroenterol. 2022 Apr;15(2):310-319. doi: 10.1007/s12328-022-01600-0. Epub 2022 Feb 8. PMID 35133625